CLINICAL TRIAL: NCT03336671
Title: Management of Pediatric Chronic Rhinosinusitis in Asthmatic Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1009628
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Chronic Sinusitis; Adenoid Disease - Chronic
Keywords: Pediatric; Chronic Sinusitis
MeSH Terms: interventions — Adenoidectomy

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenoidectomy (Active Comparator): Current standard of care for pediatric chronic rhino sinusitis.
  Interventions: Procedure: Adenoidectomy
- Adenoidectomy plus Endoscopic Sinus Surgery (Experimental): endoscopic sinus surgery in addition to adenoidectomy
  Interventions: Procedure: Endoscopic Sinus surgery; Procedure: Adenoidectomy

INTERVENTIONS:
Procedure: Endoscopic Sinus surgery — Endoscopic sinus surgery would be tailored to abnormal findings in the CT scan, as is the standard of care. Radiologists typically examine sinonasal disease of the sinuses, and they would also be requested to comment on the patency of the osteo-meatal unit, as this is a component of the Lund-McKay score. The Lund-McKay score is an objective radiologic grade of the severity of sinusitis. If there is sinus thickening, or narrowing of the OMU, endoscopic sinus surgery would be tailored to this using either balloon sinuplasty or traditional antrostomy. Patient undergoing endoscopic sinus surgery will likely have at least a maxillary antrostomy and anterior ethmoidectomy performed, with frontal sinusotomy, posterior ethmoidectomy, and sphenoidotomy performed depending on CT or endoscopy findings.
  Other Names: Functional Endoscopic Sinus Surgery
  Arms: Adenoidectomy plus Endoscopic Sinus Surgery
Procedure: Adenoidectomy — Adenoidectomy performed, routine, as a singular procedure not combined with any sinus surgery.

SUMMARY:
The objectives of this study would be to determine the most effective management for pediatric patients with chronic rhinosinusitis and asthma who fail medical management. The Sinus and Nasal Quality of Life Survey (SN-5), a validated tool, will be used to track symptoms of pediatric chronic rhinosinusitis. A decrease in at least 0.5 is felt to represent an improvement in symptom control. In this study, the SN-5 at one year post intervention will be the primary endpoint. Secondary endpoints include complications, revision surgery, and post operative endoscopy scores.

DETAILED DESCRIPTION:
Indications for surgery for pediatric chronic rhinosinusitis currently lacks scientific consensus. In general, children who fail medical management are candidates for surgery. Currently, pre-operative evaluation with a CT scan of the sinuses is the gold standard prior to sinus surgery. However, the role of the adenoids and adenoiditis in pediatric chronic sinusitis is incompletely understood. Adenoids may contribute to sinusitis both as a bacterial reservoir and obstruct nasal secretion drainage, owing to their larger relative size in children. Adenoidectomy alone has been found to improve symptoms in 75% of children.

It has been found that 50% of children continued to be symptomatic after adenoidectomy, and went on to require endoscopic sinus surgery (ESS). In addition, of the group that failed, 58% had asthma. Overall, asthma and age have been the only known risk factors for failure of adenoidectomy.

Specific Objectives The objectives of this study would be to determine the most effective management for pediatric patients with chronic rhinosinusitis and asthma who fail medical management. Outcomes will be evaluated using the SN-5, a validated tool used to track symptoms of pediatric chronic rhinosinusitis. A decrease in at least 0.5 is felt to represent an improvement in symptom control. In this study, the SN-5 at one year post intervention will be the primary endpoint. Secondary endpoints include complications, revision surgery, and post operative endoscopy scores.

Study Design

The primary outcome is the SN-5 score one year post surgery. A change of 0.5-1.0 is considered a mild improvement, while a change of at least 1.0 is considered a moderate improvement.

Sixty patients are required to have an 80% chance of detecting, as significant at the 5% level, an increase in the primary outcome measure from 47% in the control group to 80% in the experimental group.

Statistical Methods:

Univariate statistical analysis using chi-square in analysis of binary outcomes. In addition paired t test of preoperative and postoperative SN-5 scores will be performed.

Data Analysis and Interpretation:

Analysis of SN-5, and comparison of Lund-McKay(CT) scores along with post operative endoscopy Kennedy scores.

Study Procedures:

The patient's will initially be seen as a referral to the otolaryngology clinic for symptoms including chronic rhinosinusitis. If they meet inclusion criteria, they will be offered enrollment into the study and consent will be obtained. Their symptoms will be followed at each visit with the SN-5, a validated symptom-scoring tool to evaluate pediatric chronic rhinosinusitis.

If the patient does not improve with medical therapy alone after review of the SN-5 and in discussion with caregivers, he or she will be offered entry into the study, with consent, CT scan of the sinuses, and will be randomized to two different treatment arms. The first is adenoidectomy. The patient will then be followed at defined intervals with evaluation of symptoms by SN-5. Should symptoms worsen or not improve, they will then be offered endoscopic sinus surgery, with findings from the CT scan of the sinuses to guide operative intervention. Adenoidectomy followed by endoscopic sinus surgery is the current standard of care and serves as the control arm. In the other experimental or study arm, the patient will undergo adenoidectomy with endoscopic sinus surgery at the same time. Radioallergosorbent test blood testing for allergies would be performed at the time of surgery in both groups.

For patients who initially improve with medical therapy, but relapse at a later time, they may either undergo consent and randomization if they relapse within a year or a repeat course of medical therapy if it has been one year since previous medical therapy.

Endoscopic sinus surgery, in both arms would be tailored to abnormal findings in the CT scan, as is the standard of care. Radiologists typically examine sinonasal disease of the sinuses, and they would also be requested to comment on the patency of the osteo-meatal unit, as this is a component of the Lund-McKay score. The Lund-McKay score is an objective radiologic grade of the severity of sinusitis. If there is sinus thickening, or narrowing of the osteomeatal unit, endoscopic sinus surgery would be tailored to this using either balloon sinus opening or traditional antrostomy. Patient undergoing endoscopic sinus surgery will likely have at least a maxillary antrostomy and anterior ethmoidectomy performed, with frontal sinusotomy, posterior ethmoidectomy, and sphenoidotomy performed depending on CT or endoscopy findings.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-12 at time of study enrollment.
2. Presence of chronic sinusitis: >90 days 2 or more symptoms of purulent rhinorrhea, nasal obstruction, facial pressure/pain, or cough
3. Presence of asthma, as documented in the medical record by the patient's pediatrician and/or pulmonologist
4. Failure of medical management of pediatric chronic rhinosinusitis, which current guidelines recommend extended empiric antibiotics for 21 days, which will be either Augmentin or clindamycin in penicillin allergic patients, at standard pediatric weight based dosing. In addition, Flonase nasal spray and nasal saline treatment for three weeks. Failure is considered persistent symptoms despite treatment with the above within the past year.

Exclusion Criteria:

1. Previous sinus surgery,
2. Previous adenoidectomy, or
3. Presence of cystic fibrosis,
4. Presence of antrochoanal polyp,
5. Immunodeficiency
6. Fungal infection.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
SN-5 at one year post procedure | One year
  A validated tool used to track symptoms of pediatric chronic rhinosinusitis, improvement greater than 0.5

SECONDARY OUTCOMES:
Revision/Alternate procedure, endoscopic sinus surgery | Two Years
  Requirement of the alternate procedure or a revision procedure.
Antibiotic use after surgical procedure | Two years
  Relapse of chronic rhinosinusitis, if treated with antibiotics will be documented as the number of courses of antibiotics taken for rhino sinusitis in two years after the initial procedure
Complication Rate | Two Years
  Complications associated with medical management, or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haidy Marzouk, MD, Principal Investigator — State University of New York - Upstate Medical University; Mark Arnold, MD, Study Director — 315 464-4678
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No